CLINICAL TRIAL: NCT00004851
Title: Generation of Anti-HCV Antibodies From Bone Marrow: Defining the Repertoire of Immune Response to HCV Quasispecies
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990090; 99-CC-0090
Record Dates: First submitted 2000-03-02; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-03

CONDITIONS: Hepatitis C
Keywords: HCV Antibody Library
MeSH Terms: conditions — Hepatitis C

SUMMARY:
To generate a library of genes that reflect the entirety of antibody responses to hepatitis C virus (HCV) made during the 20-year course of HCV infection in a single patient (WH) whose viral quasispecies has been extensively characterized. In addition to characterizing the sequential events in antibody formation and their relationship to the changing pattern of viral quasispecies, we hope to identify neutralizing antibodies and the epitopes to which they are directed. Ultimately we seek to gain insight into the host mechanisms that suppress viral replication and to translate this to therapeutic and preventive modalities.

DETAILED DESCRIPTION:
To generate a library of genes that reflect the entirety of antibody responses to hepatitis C virus (HCV) made during the 20-year course of HCV infection in a single patient (WH) whose viral quasispecies has been extensively characterized. In addition to characterizing the sequential events in antibody formation and their relationship to the changing pattern of viral quasispecies, we hope to identify neutralizing antibodies and the epitopes to which they are directed. Ultimately we seek to gain insight into the host mechanisms that suppress viral replication and to translate this to therapeutic and preventive modalities.

ELIGIBILITY:
Persistent infection with mild hepatitis that is non-progressive.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1
Dates: Start 1999-04; Study Completion 2001-05

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Feinstone SM, Alter HJ, Dienes HP, Shimizu Y, Popper H, Blackmore D, Sly D, London WT, Purcell RH. Non-A, non-B hepatitis in chimpanzees and marmosets. J Infect Dis. 1981 Dec;144(6):588-98. doi: 10.1093/infdis/144.6.588. PMID 6799586
- [Background] Hijikata M, Shimizu YK, Kato H, Iwamoto A, Shih JW, Alter HJ, Purcell RH, Yoshikura H. Equilibrium centrifugation studies of hepatitis C virus: evidence for circulating immune complexes. J Virol. 1993 Apr;67(4):1953-8. doi: 10.1128/JVI.67.4.1953-1958.1993. PMID 8383220
- [Background] Shimizu YK, Hijikata M, Iwamoto A, Alter HJ, Purcell RH, Yoshikura H. Neutralizing antibodies against hepatitis C virus and the emergence of neutralization escape mutant viruses. J Virol. 1994 Mar;68(3):1494-500. doi: 10.1128/JVI.68.3.1494-1500.1994. PMID 8107212